CLINICAL TRIAL: NCT04930575
Title: Muscle Energy Technique Versus Mulligan Technique for Treating Neck Pain in Breast Feeding Women
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Heba Mohamed Mohamed Mohamed El-Basiony, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HElbasiony_MSc
Record Dates: First submitted 2021-06-11; First posted 2021-06-18 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-06

CONDITIONS: Neck Pain; Breast Feeding
MeSH Terms: conditions — Neck Pain; Breast Feeding

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Muscle Energy Technique group (Experimental): Patients in the group (B) will receive muscle energy technique on tonic muscles in the neck (sternocleidomastoid, scalenes, levator scapulae, and upper trapezius) in addition to strengthening exercise for deep cervical flexors and advice to correct positions three times per week for 4 weeks.
  The aim of the Muscle Energy Technique in the context of NP is to decrease pain, improve movement, motor control, and function and thereby reduce disability.
  A biomechanical correction approach can lead to the normalization of spinal curvatures and a decrease in the compressional and tensional stress on joints and soft tissues of the body thus alleviating the patient's signs and symptoms.
  Interventions: Other: Muscle Energy Technique
- Mulligan Technique group (Experimental): Patient in group A will receive specialized SNAGs technique adapted from Mulligan (2005), in addition to strengthening exercise for DNF muscles and advice to correct position three times per week for 4 weeks.
  Interventions: Other: Mulligan Technique

INTERVENTIONS:
Other: Muscle Energy Technique — A biomechanical correction approach can lead to the normalization of spinal curvatures and a decrease in the compressional and tensional stress on joints and soft tissues of the body.
  Arms: Muscle Energy Technique group
Other: Mulligan Technique — * The patient will be in a supportive low back chair, thus cervical region will be in a vertical position (Weight-bearing position) with the therapist position will be behind the patient.
  * Then the therapist will move the spinous process up in the direction that must follow the apophyseal joint plane under treatment, that is, toward the eye ball. While sustaining this pain-free accessory glide, the patient will be instructed to actively perform the physiological movement gradually until the end ROM with over pressure at the end of the range.
  Arms: Mulligan Technique group

SUMMARY:
The purpose of this study will determine the effect of muscle energy technique versus mulligan technique on neck pain in breastfeeding women.

DETAILED DESCRIPTION:
Conservative treatments used to manage neck pain are numerous and include usual medical care ( face to face interview, education, reassurance, medication, ergonomic and stay active advice), various forms of exercise, massage, and acupuncture among others, but a lack of evidence regarding their relative efficacy was found.

More research is needed to determine specific exercise programs that can decrease neck pain in breastfeeding women. So, this study will be conducted to determine clinical evidence of the effectiveness of muscle energy technique versus mulligan technique on neck pain, which constituted a great problem facing the mother during the breastfeeding period.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be examined by a physician before the study and will be chosen according to the following criteria:
* All patients will be in the breastfeeding period at least 6 weeks after delivery.
* All patients will be clinically diagnosed with neck pain (with no neurological or rheumatological problem).
* Their ages will range from 25-35years.
* Their BMI will be less than 30 kg/m².
* Their parity will not be more than 3 times.

Exclusion Criteria:

* The patients will be excluded if they have any of the followings:

  1. Any contraindication to spinal mobilization (e.g., inflammation, infection, advanced degeneration, congenital malformation, trauma, cerebrovascular abnormalities).
  2. Positive neurological examination (presence of positive motor reflex, or sensory abnormalities indicating spinal root compression).
  3. Cervical spine surgery or stenosis, metabolic or systemic disorder, or cancer.
  4. Associated pathology of the upper cervical region or upper limb that may cause overlapping with the clinical finding as referred pain from the costotransverse joint, rotator cuff tendonitis, and cervical rib syndrome.

Ages: 25 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Breast feeding women
Enrollment: 32 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-06-15 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Assessing the change in Cervical pain level | Baseline and 4 weeks post-intervention
  Assessment via using Visual Analogue Scale that continuous data analysis and uses a 10 cm long with 0 (no pain) and 10 (worst pain). Patient will be asked to place a mark along the line to denote their level of pain.
Assessing the change in Functional disability | Baseline and 4 weeks post-intervention
  Assessment via using Neck pain disability index questionnaire consists of 10 items each of them is scored from 0 to 5. The total maximum score is therefore 50.The original report provided scoring interval for interpretation, as; (0-4) = no disability, (5-14) mild, (15-24) moderate, (25-34) sever, (above34) complete disability.
Assessing the change in Cervical Range Of Motion | Baseline and 4 weeks post-intervention
  Assessment via using Digital goniometer is valid and has good reliability for measuring cervical spine range of motion.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Physical Therapy Cairo University, Dokki, Egypt

IPD SHARING:
Plan to Share IPD: No